CLINICAL TRIAL: NCT05172011
Title: NIH RECOVER: A Multi-site Observational Study of Post-acute Sequalae of SARS-CoV-2 Infection in Children
Brief Title: Understanding the Long-term Impact of COVID on Children and Families
Status: Active, not recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 21-01231
Record Dates: First submitted 2021-12-27; First posted 2021-12-29 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: SARS-CoV-2 Infection
Keywords: Post Acute Sequalae of SARS-CoV-2 (PASC)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Tier 1: Saliva and blood, Tier 2: Blood and urine, Tier 3: Blood, sputum, nasal swab, oral swab, skin swab, stool, urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Extant, Clinical and De Novo Cohort -- INFECTED: SARS-CoV-2 infected children and young adults with and without current or prior PASC-like symptoms, including infected individuals with history of multisystem inflammatory syndrome in children (MIS-C), and infants born in the context of maternal SARS-CoV-2 infection during pregnancy
- Extant, Clinical and De Novo Cohort -- UNINFECTED: SARS-CoV-2 uninfected children and infants born to uninfected mothers
- Acute Cohort -- INFECTED: Newly SARS-CoV-2 infected individuals (≤4 weeks since onset of symptoms or positive laboratory testing)
- Acute Cohort -- UNINFECTED: Contemporaneous SARS-CoV-2 uninfected individuals selected from the same population as newly SARS-CoV-2 infected individuals
- Post-acute cohort -- INFECTED: Post-acute infected individuals (>4 weeks after initial symptoms or positive laboratory testing) in the extant, clinical and de novo cohorts, including infants born in the context of maternal SARS-CoV-2 infection during pregnancy, will be enrolled 1-24 months after initial SARS-CoV-2 infection.
- Post-acute cohort -- UNINFECTED: Uninfected individuals will be derived from a similar population with respect to age, sex, race and ethnicity, geographic origin, sociodemographics, and time of enrollment as the infected individuals.
- Post-COVID Vaccine Myocarditis: Individuals with history of myocarditis after receiving COVID-19 vaccine.
- Primary Caregivers: The primary caregiver of the child or young adult may optionally participate in the study.
- Biological Parent: If the primary caregiver is a biological parent, the other biological parent may optionally participate in the study

SUMMARY:
This is a combined retrospective and prospective, longitudinal, observational meta-cohort of individuals age 0-25 years who will enter the cohort with and without SARS-CoV-2 infection at varying stages before and after infection. Individuals with and without SARS-CoV-2 infection and with or without PASC symptoms will be followed to identify risk factors and occurrence of PASC. This study will be conducted in the United States and participants will be recruited through inpatient, outpatient, and community-based settings. Study data including age, demographics, social determinants of health, medical history, vaccination history, details of acute SARS-CoV-2 infection, overall health and physical function, and PASC symptoms will be reported by participants or collected from the electronic health record using a case report form at specified intervals. Biologic specimens will be collected at specified intervals, with some tests performed in local clinical laboratories and others performed by centralized research centers or banked in the Biospecimen Repository. Advanced clinical examinations and radiologic examinations will be performed at local study sites with cross-site standardization.

DETAILED DESCRIPTION:
Ambidirectional longitudinal meta-cohort study (combined retrospective and prospective) with nested case-control studies.

ELIGIBILITY:
Inclusion Criteria:

Infected Cohort:

Patients will be eligible for inclusion according to the following criteria:

1. Ages newborn-25 years
2. Infected individuals will have suspected, probable, or confirmed SARS-CoV-2 infection as defined by WHO criteria within 24 months of enrollment or have been born to a mother meeting these criteria during pregnancy (congenitally exposed)
3. Children/young adults with or without history of MIS-C are eligible
4. Children/young adults with or without history of SARS-CoV-2 vaccination are eligible
5. Children/young adults with evidence of past SARS-CoV-2 infection based on serum antibody profile are eligible (with or without history of acute symptoms)
6. Children/young adults with recurrent SARS-CoV-2 infections and those with post-vaccination (breakthrough) infections are eligible to participate
7. Participants are eligible without exclusion related to sex, race/ethnicity, geography, nationality, severity of disease, or underlying health conditions

Children/Young Adults with Suspected SARS-Cov-2 Infection

Children/young adults who meet these clinical criteria:

At least one of these clinical criteria:

* Acute onset of fever and cough OR
* Acute onset of ANY THREE OR MORE of the following signs or symptoms: fever, cough, general weakness /fatigue, headache, myalgia, sore throat, coryza, dyspnea, anorexia/nausea/vomiting, diarrhea, altered mental status.

AND at least one of these epidemiological criteria:

1. Residing or working in an area with a high risk of transmission of virus: closed residential, school or camp settings anytime within the 14 days before symptom onset; OR
2. Residing or travel to an area with community transmission anytime within the 14 days before symptom onset; OR
3. Any known household contact or any member of the household working in any health care setting, including within health facilities or within the community; anytime within the 14 days before symptom onset.
4. A patient with history of severe acute respiratory illness (SARI):

   - SARI: acute respiratory infection with history of fever or measured fever of ≥ 38 C°; and cough; with onset within the last 10 days; and requires hospitalization
5. An asymptomatic person not meeting epidemiologic criteria with a positive SARS-CoV-2 Antigen-RDT.

Children/Young Adults with Probable SARS-Cov-2 Infection

1. A patient who meets clinical criteria above AND is a contact of a probable or confirmed case or linked to a COVID-19 cluster; OR
2. A suspect case with chest imaging showing findings suggestive of COVID-19 disease; OR
3. A person with recent onset of anosmia (loss of smell) or ageusia (loss of taste) in the absence of any other identified cause

Children/Young Adults with Confirmed SARS-Cov-2 Infection

1. A person with a positive Nucleic Acid Amplification Test (NAAT); OR
2. A person with a positive SARS-CoV-2Antigen-RDT AND meeting either the probable case definition or suspect criteria A OR B; OR
3. An asymptomatic person with a positive SARS-CoV-2 Antigen-RDT who is a contact of a probable or confirmed case

Children/Young Adults with Asymptomatic SARS-CoV-2 Infection

1. A person without history of acute COVID-19 symptoms who has one or more of the epidemiological exposures for suspected infection and who also meets criteria b or c for suspected or probable infection, or who meets any of the criteria for confirmed infection
2. A person without history of acute COVID-19 symptoms who has positive nucleocapsid antibody test result in medical history or Tier 1 testing with or without NAAT or RDT testing or known contact to a probable or confirmed case.

Non-Infected Cohort

A person who meets the following criteria will qualify for enrollment as a non-infected control subject:

1. Does not meet WHO criteria for a suspected, probable, or confirmed case of SARS-CoV-2 infection AND
2. Does not have serological evidence of past asymptomatic SARS-CoV-2 infection in medical history or Tier 1 testing, AND
3. Lives in the same communities or recruited from the same sources as those in the SARS-CoV-2 infected cohort, AND
4. Either not hospitalized for any reason in prior 3 months, or hospitalized (with or without ICU stay) within the prior 3 months
5. Uninfected individuals may participate independent of their vaccination status
6. Uninfected individuals who develop SARS-CoV-2 infection during the study period will be reassigned to the SARS-Cov-2 infected group and will be considered to have been enrolled prior to SARS-CoV-2 infection.

Children (≤3 years of age) born in and out of the context of maternal SARS-CoV-2 infection during pregnancy.

1. Children ≤3 years of age born to a childbearing parent with history of suspected, probable, or confirmed SARS-COV-2 infection during pregnancy (according the same criteria listed for the infected child cohort) will be enrolled in the study from existing research cohorts at the maternal fetal medicine sites in the RECOVER. network.
2. Children ≤3 years of age born to a childbearing parent without history of SARS-COV-2 infection during pregnancy (according to the same criteria listed for the non-infected child cohort) will also be enrolled from the same existing research cohorts at maternal fetal medicine sites in the RECOVER network.

Children with MIS-C

Children/young adults with SARS-CoV-2 infection who have history of MIS-C meeting the CDC definition:

1. An individual aged <21 years presenting with fever*, laboratory evidence of inflammation**, and evidence of clinically severe illness requiring hospitalization, with multisystem (>2) organ involvement (cardiac, renal, respiratory, hematologic, gastrointestinal, dermatologic or neurological); AND
2. No alternative plausible diagnoses; AND
3. Positive for current or recent SARS-CoV-2 infection by RT-PCR, serology, or antigen test; or exposure to a suspected or confirmed COVID-19 case within the 4 weeks prior to the onset of symptoms.

   * Fever >38.0°C for ≥24 hours, or report of subjective fever lasting ≥24 hours **Including, but not limited to, one or more of the following: an elevated C-reactive protein (CRP), erythrocyte sedimentation rate (ESR), fibrinogen, procalcitonin, d-dimer, ferritin, lactic acid dehydrogenase (LDH), or interleukin 6 (IL-6), elevated neutrophils, reduced lymphocytes and low albumin Young adults with past history of MIS-C with current ages 22-25 years are eligible to participate.

Children/Young Adults with Post-Vaccine Myocarditis

1. Age 3-25 years
2. Recipient of mRNA COVID-19 vaccination within last 4 weeks
3. Children or young adults with or without history of SARS-CoV-2 infection are eligible
4. Children or young adults with or without history of MIS-C are eligible (if any prior MIS-C-related cardiac abnormalities are known to have resolved pre-vaccination)
5. No other known auto-immune or other immune dysregulation disease
6. Participants are eligible without exclusion related to sex, race/ethnicity, geography, nationality, severity of disease, or underlying health conditions
7. Clinical evidence of probable or confirmed myocarditis based on the following criteria:

Children and young adults ages 3-25 years with presence of ≥1 new or worsening of the following clinical symptoms:

* chest pain, pressure, or discomfort
* dyspnea, shortness of breath, or pain with breathing
* palpitations
* syncope

OR, children aged 3-12 years might instead have ≥2 of the following symptoms:

* irritability
* vomiting
* poor feeding
* tachypnea
* lethargy AND

  ≥1 new finding of:
* troponin level above upper limit of normal (any type of troponin)
* abnormal electrocardiogram (ECG or EKG) or rhythm monitoring findings consistent with myocarditis
* abnormal cardiac function or wall motion abnormalities on echocardiogram
* cardiac MRI findings consistent with myocarditis
* histopathologic confirmation of myocarditis (Definite myocarditis)¶ AND
* No other identifiable cause of the symptoms and finding

Entry criteria are adapted from the CDC definition based on the assumptions that COVID-19 vaccines will be available in the future to children <5 years of age.

Primary Caregiver Entry Criteria

1. A primary caregiver is defined as an individual, such as a family member (biological or nonbiological) or legal guardian, who is responsible for the care of the enrolled child and resides in the same household as the child. When possible, the primary caregiver identified at study entry will remain in the same role throughout the study.
2. The primary caregiver is the caregiver who spends the most time with the child or young adult, has substantial responsibility for taking care of him/her on a daily basis, and is most knowledgeable about him/her.
3. If two or more persons share equally in the caregiver responsibilities for the child or young adult, the person selected by the family to fill out study forms both about themselves and the child will be considered the primary caregiver.
4. If a biological family member primary caregiver has not reached the legal age of majority in their jurisdiction, the parent/legal guardian for the minor primary caregiver will provide consent for participation, with assent provided by the minor caregiver.
5. A nonbiological primary caregiver or legal guardian serving as primary caregiver must be above the legal age of majority in their jurisdiction.
6. The primary caregiver cannot be a babysitter or other childcare provider who receives money to care for the child.

Biological Parent Entry Criteria

- If the primary caregiver is a biological parent of the child or young adult who is participating in the study, the other biological parent may be enrolled to provide a home sample of saliva for DNA analysis.

Exclusion Criteria

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Any child, young adult, caregiver, or other biological parent who in the opinion of the site investigator may be at increased risk of adverse events during participation in the study, or who may not be able to complete study procedures due to co-morbid disease or disability.
2. Any young adult age above the age of majority who lacks capacity to provide consent
3. Nonviable neonates and neonates of uncertain viability as determined by the treating physician
4. Any child, young, adult, or caregiver with co-morbid illness with expected survival <2 years
5. Any child who is being given up for adoption or is a ward of the state
6. Any caregiver or other biological parent who is incarcerated, or who lacks capacity to provide consent
7. Currently enrolled in the study Understanding the Long-term Impact of COVID-19 in Adults

Max Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Infected: Individuals less than 25 years of age meeting WHO criteria for suspected, probable or confirmed SARS-CoV-2 infection on or after March 1, 2020; or those born to a mother meeting these criteria during pregnancy.
  Uninfected: Individuals less than 25 years of age who have never met any of the WHO criteria for suspected, probable or confirmed SARS-CoV-2 infection.
Sampling Method: Non-Probability Sample
Enrollment: 15028 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-05-23 (Estimated)

PRIMARY OUTCOMES:
Caregiver SARS-CoV-2 Infection Status | Baseline
  Initial SARS-CoV-2 infection is reported via remote patient report (electronic, paper or telephone assessments) and EHR. Infection categories include: SARS CoV 2 PCR result, SARS CoV 2 antigen result, SARS CoV 2 antibody result, SARS CoV 2 sequencing performed, diagnosed by a doctor based on symptoms, suspected by participant but not diagnosed by a doctor.
Child SARS-CoV-2 Infection Status | Baseline
  Initial SARS-CoV-2 infection is reported via remote patient report (electronic, paper or telephone assessments) and EHR. Infection categories include: SARS CoV 2 PCR result, SARS CoV 2 antigen result, SARS CoV 2 antibody result, SARS CoV 2 sequencing performed, diagnosed by a doctor based on symptoms, suspected by participant but not diagnosed by a doctor.
Caregiver Severity of SARS-CoV-2 Infection | Baseline
  Severity levels are reported via remote patient report (electronic, paper or telephone assessments) and EHR. NIH severity levels include: asymptomatic or presymptomatic, mild illness, moderate illness, severe illness, and critical illness.
Child Severity of SARS-CoV-2 Infection | Baseline
  Severity levels are reported via remote patient report (electronic, paper or telephone assessments) and EHR. NIH severity levels include: asymptomatic or presymptomatic, mild illness, moderate illness, severe illness, and critical illness.
Caregiver Previous In-Hospital SARS-CoV-2 Treatment Record | Baseline
  Treatments will be reported via remote patient report (electronic, paper, or telephone assessment) and EHR -- Treated with corticosteroids , Treated with hydroxychloroquine, Treated with lopinavir, ritonavir, other antiviral, Treated with monoclonal antibody, Treated with therapeutic anticoagulation, Treated with antibiotics.
Child Previous In-Hospital SARS-CoV-2 Treatment Record | Baseline
  Treatments will be reported via remote patient report (electronic, paper, or telephone assessment) and EHR -- Treated with corticosteroids , Treated with hydroxychloroquine, Treated with lopinavir, ritonavir, other antiviral, Treated with monoclonal antibody, Treated with therapeutic anticoagulation, Treated with antibiotics.
Caregiver Symptoms | Baseline, up to Month 48
  Symptoms will be reported via remote patient report, in-person patient report, or EHR
Child Symptoms | Baseline, up to Month 48
  Symptoms will be reported via remote patient report, in-person patient report, or EHR -- symptoms include: Nasal Congestion, Trouble breathing, Pain when breathing, Chest pain, Palpitations/heart racing, Dizziness/lightheadedness, Fainting, Change in hearing/ringing in ears, Blurred vision, Change in smell, Change in taste, Problems with teeth or gums, Tremors/shakiness, Feeling off-balance or unsteady, Feeling tingling or "pins and needles", Seizures/fits, Muscle weakness, Difficulty sleeping, Excessive sleepiness, Fatigue/Low energy, Feeling exhausted after walking, Poor appetite, Stomach pains/cramps, Nausea, Vomiting, Diarrhea, Constipation, Problems with urination, Skin rash, Problems with memory, Problems with concentration, Speech difficulty, Anxiety, Depression, Body pain, Headache, Problems swallowing or chewing, Change in menstruation
Caregiver SARS-CoV-2 Vaccination Status | Baseline, up to Month 48
  Vaccination in status will be reported via remote patient report, in-person patient report, or EHR.
Change in Child SARS-CoV-2 Vaccination Status | Week 8, up to Month 48
  Vaccination in status will be reported via remote patient report, in-person patient report, or EHR.
Change in Caregiver SARS-CoV-2 Treatment Record | Month 12, up to Month 48
  Treatments will be reported via remote patient report, in-person patient report, or EHR -- Treated with corticosteroids, Treated with hydroxychloroquine, Treated with lopinavir, ritonavir, other antiviral, Treated with monoclonal antibody, Treated with therapeutic anticoagulation, Treated with antibiotics.
Change in Child SARS-CoV-2 Treatment Record | Week 8, up to Month 48
  Treatments will be reported via remote patient report, in-person patient report, or EHR -- Treated with corticosteroids, Treated with hydroxychloroquine, Treated with lopinavir, ritonavir, other antiviral, Treated with monoclonal antibody, Treated with therapeutic anticoagulation, Treated with antibiotics.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Katz, MD, MS, Principal Investigator — NYU Langone Health; Andrea Troxel, ScD, Principal Investigator — NYU Langone Health; Leora Horwitz, MD, Principal Investigator — NYU Langone Health
Locations (65):
- United States (65):
  - University of Alabama at Birmingham (Pregnancy Cohort), Birmingham, Alabama
  - Arkansas Children's Hospital and Research Institute, Little Rock, Arkansas
  - University of California San Diego, La Jolla, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California San Diego Health - Rady Children's Hospital, San Diego, California
  - University of California San Francisco (Pregnancy Cohort), San Francisco, California
  - University of California San Francisco, San Francisco, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale School of Medicine (YSM), New Haven, Connecticut
  - ChristianaCare Health System, Newark, Delaware
  - Nemours Children's Health, Wilmington, Delaware
  - George Washington University, Washington D.C., District of Columbia
  - Kapi'olani Medical Center for Women & Children, Honolulu, Hawaii
  - Northwestern University, Evanston, Illinois
  - Northshore University HealthSystem, Glenview, Illinois
  - American Academy of Pediatrics, Itasca, Illinois
  - American Academy of Family Physicians, Leawood, Kansas
  - University of Louisville - Norton Children's Hospital, Louisville, Kentucky
  - Louisiana State University (LSU) - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Tulane University, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Mass General Brigham - Harvard University, Boston, Massachusetts
  - Harvard Medical School, Boston, Massachusetts
  - Harvard School Of Public Health, Boston, Massachusetts
  - Northeastern University, Boston, Massachusetts
  - Central Michigan University - College of Medicine, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University Of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth-Hitchcock, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers University, New Brunswick, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - The Pediatric Specialty Center at Saint Barnabas, West Orange, New Jersey
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - NYU Langone Health, New York, New York
  - Columbia University, New York, New York
  - Columbia University (Pregnancy), New York, New York
  - NewYork-Presbyterian Hospital, Queens, New York
  - New York Medical College, Valhalla, New York
  - University of North Carolina (UNC) at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - WakeMed Health & Hospitals, Raleigh, North Carolina
  - Good Samaritan Hospital, Cincinnati, Ohio
  - University Hospitals MacDonald's Women's Hospital, Cleveland, Ohio
  - Metrohealth System, Cleveland, Ohio
  - The MetroHealth System (Pregnancy Cohort), Cleveland, Ohio
  - The Ohio State University - Wexner Medical Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Children's Mercy Hospital, Fairfield, Ohio
  - University of Oklahoma Health Sciences Center (OUHSC), Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Women & Infants Hospital, Providence, Rhode Island
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Prisma Health Upstate, Greenville, South Carolina
  - Avera Research Institute, Sioux Falls, South Dakota
  - University of Texas Medical Branch (UTMB) Galveston, Galveston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Utah Health, Salt Lake City, Utah
  - University of Vermont (UVM) Children's Hospital, Burlington, Vermont
  - Virginia Commonwealth University, Richmond, Virginia
  - West Virginia University, Morgantown, West Virginia
  - Medical College Of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available beginning 9 months with no end date.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to RECOVER_CSC@NYULangone.org To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Gross RS, Thaweethai T, Rosenzweig EB, Chan J, Chibnik LB, Cicek MS, Elliott AJ, Flaherman VJ, Foulkes AS, Gage Witvliet M, Gallagher R, Gennaro ML, Jernigan TL, Karlson EW, Katz SD, Kinser PA, Kleinman LC, Lamendola-Essel MF, Milner JD, Mohandas S, Mudumbi PC, Newburger JW, Rhee KE, Salisbury AL, Snowden JN, Stein CR, Stockwell MS, Tantisira KG, Thomason ME, Truong DT, Warburton D, Wood JC, Ahmed S, Akerlundh A, Alshawabkeh AN, Anderson BR, Aschner JL, Atz AM, Aupperle RL, Baker FC, Balaraman V, Banerjee D, Barch DM, Baskin-Sommers A, Bhuiyan S, Bind MC, Bogie AL, Bradford T, Buchbinder NC, Bueler E, Bukulmez H, Casey BJ, Chang L, Chrisant M, Clark DB, Clifton RG, Clouser KN, Cottrell L, Cowan K, D'Sa V, Dapretto M, Dasgupta S, Dehority W, Dionne A, Dummer KB, Elias MD, Esquenazi-Karonika S, Evans DN, Faustino EVS, Fiks AG, Forsha D, Foxe JJ, Friedman NP, Fry G, Gaur S, Gee DG, Gray KM, Handler S, Harahsheh AS, Hasbani K, Heath AC, Hebson C, Heitzeg MM, Hester CM, Hill S, Hobart-Porter L, Hong TKF, Horowitz CR, Hsia DS, Huentelman M, Hummel KD, Irby K, Jacobus J, Jacoby VL, Jone PN, Kaelber DC, Kasmarcak TJ, Kluko MJ, Kosut JS, Laird AR, Landeo-Gutierrez J, Lang SM, Larson CL, Lim PPC, Lisdahl KM, McCrindle BW, McCulloh RJ, McHugh K, Mendelsohn AL, Metz TD, Miller J, Mitchell EC, Morgan LM, Muller-Oehring EM, Nahin ER, Neale MC, Ness-Cochinwala M, Nolan SM, Oliveira CR, Osakwe O, Oster ME, Payne RM, Portman MA, Raissy H, Randall IG, Rao S, Reeder HT, Rosas JM, Russell MW, Sabati AA, Sanil Y, Sato AI, Schechter MS, Selvarangan R, Sexson Tejtel SK, Shakti D, Sharma K, Squeglia LM, Srivastava S, Stevenson MD, Szmuszkovicz J, Talavera-Barber MM, Teufel RJ 2nd, Thacker D, Trachtenberg F, Udosen MM, Warner MR, Watson SE, Werzberger A, Weyer JC, Wood MJ, Yin HS, Zempsky WT, Zimmerman E, Dreyer BP; RECOVER-Pediatric Consortium. Researching COVID to enhance recovery (RECOVER) pediatric study protocol: Rationale, objectives and design. PLoS One. 2024 May 7;19(5):e0285635. doi: 10.1371/journal.pone.0285635. eCollection 2024. PMID 38713673
- [Derived] Metz TD, Clifton RG, Gallagher R, Gross RS, Horwitz LI, Jacoby VL, Martin-Herz SP, Peralta-Carcelen M, Reeder HT, Beamon CJ, Chan J, Chang AA, Costantine MM, Fitzgerald ML, Foulkes AS, Gibson KS, Guthe N, Habli M, Hackney DN, Hoffman MK, Hoffman MC, Hughes BL, Katz SD, Laleau V, Mallett G, Mendez-Figueroa H, Monzon V, Palatnik A, Palomares KTS, Parry S, Pettker CM, Plunkett BA, Poppas A, Reddy UM, Rouse DJ, Saade GR, Sandoval GJ, Schlater SM, Sciurba FC, Simhan HN, Skupski DW, Sowles A, Thaweethai T, Thomas GL, Thorp JM Jr, Tita AT, Weiner SJ, Weigand S, Yee LM, Flaherman VJ; RECOVER Initiative. Researching COVID to enhance recovery (RECOVER) pregnancy study: Rationale, objectives and design. PLoS One. 2023 Dec 21;18(12):e0285351. doi: 10.1371/journal.pone.0285351. eCollection 2023. PMID 38128008
- [Derived] Gross R, Thaweethai T, Rosenzweig EB, Chan J, Chibnik LB, Cicek MS, Elliott AJ, Flaherman VJ, Foulkes AS, Witvliet MG, Gallagher R, Gennaro ML, Jernigan TL, Karlson EW, Katz SD, Kinser PA, Kleinman LC, Lamendola-Essel MF, Milner JD, Mohandas S, Mudumbi PC, Newburger JW, Rhee KE, Salisbury AL, Snowden JN, Stein CR, Stockwell MS, Tantisira KG, Thomason ME, Truong DT, Warburton D, Wood JC, Ahmed S, Akerlundh A, Alshawabkeh AN, Anderson BR, Aschner JL, Atz AM, Aupperle RL, Baker FC, Balaraman V, Banerjee D, Barch DM, Baskin-Sommers A, Bhuiyan S, Bind MC, Bogie AL, Buchbinder NC, Bueler E, Bukulmez H, Casey BJ, Chang L, Clark DB, Clifton RG, Clouser KN, Cottrell L, Cowan K, D'Sa V, Dapretto M, Dasgupta S, Dehority W, Dummer KB, Elias MD, Esquenazi-Karonika S, Evans DN, Faustino EVS, Fiks AG, Forsha D, Foxe JJ, Friedman NP, Fry G, Gaur S, Gee DG, Gray KM, Harahsheh AS, Heath AC, Heitzeg MM, Hester CM, Hill S, Hobart-Porter L, Hong TKF, Horowitz CR, Hsia DS, Huentelman M, Hummel KD, Iacono WG, Irby K, Jacobus J, Jacoby VL, Jone PN, Kaelber DC, Kasmarcak TJ, Kluko MJ, Kosut JS, Laird AR, Landeo-Gutierrez J, Lang SM, Larson CL, Lim PPC, Lisdahl KM, McCrindle BW, McCulloh RJ, Mendelsohn AL, Metz TD, Morgan LM, Muller-Oehring EM, Nahin ER, Neale MC, Ness-Cochinwala M, Nolan SM, Oliveira CR, Oster ME, Payne RM, Raissy H, Randall IG, Rao S, Reeder HT, Rosas JM, Russell MW, Sabati AA, Sanil Y, Sato AI, Schechter MS, Selvarangan R, Shakti D, Sharma K, Squeglia LM, Stevenson MD, Szmuszkovicz J, Talavera-Barber MM, Teufel RJ 2nd, Thacker D, Udosen MM, Warner MR, Watson SE, Werzberger A, Weyer JC, Wood MJ, Yin HS, Zempsky WT, Zimmerman E, Dreyer BP. Researching COVID to enhance recovery (RECOVER) pediatric study protocol: Rationale, objectives and design. medRxiv [Preprint]. 2023 May 12:2023.04.27.23289228. doi: 10.1101/2023.04.27.23289228. PMID 37214806

DOCUMENTS (1):
  • Informed Consent Form (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT05172011/ICF_000.pdf